CLINICAL TRIAL: NCT01724580
Title: Compassionate Use Treatment Protocol I4V-MC-JAGA: Treatment of Conditions Expected to Benefit From JAK 1/2 Inhibition: CANDLE, CANDLE-Related Conditions, SAVI and Severe Juvenile Dermatomyositis
Brief Title: Compassionate Use Protocol for the Treatment of Autoinflammatory Syndromes
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 14559; I4V-MC-JAGA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Atypical Neutrophilic Dermatosis With Lipodystrophy and Elevated Temperature (CANDLE); Juvenile Dermatomyositis (JDM); Stimulator of Interferon Genes (STING)-Associated Vasculopathy With Onset During Infancy (SAVI); Aicardi-Goutières Syndrome (AGS)
MeSH Terms: conditions — Fever; Dermatomyositis; Bites and Stings | interventions — baricitinib

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104; INCB 028050

SUMMARY:
The Requesting Physician/Investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥17.5 months of age (or are ≥6 months of age with Aicardi-Goutières Syndrome [AGS]). Participants younger than 17.5 months of age can be considered for enrollment after discussion with the sponsor.
* Have systemic signs and symptoms of inflammation as manifested by the presence of two or more of the following symptoms: rash, fever, musculoskeletal pain, headache, fatigue, weakness, respiratory/breathing symptoms, or ulcers/ischemic lesions.
* Have an average daily Diary Score of ≥0.5 (CANDLE Diary; used also for CANDLE-related conditions, AGS Diary) or ≥1.0 (SAVI) or ≥1.0 exclusive of headache and fever symptoms (JDM Diary) assessed over at least 2 weeks prior to entry, if available. Otherwise, participants can complete the diary after study consent is signed during the screening period and meet the inclusion criteria for enrollment into the study.
* Are ≥8.5 kilogram (kg) in body weight. Participants weighing less than 8.5 kg can be considered for enrollment after discussion with the sponsor.
* Have been previously treated with at least 1 biologic therapy and, in the opinion of the investigator, did not respond or are no longer responding to therapy. If the participant has been diagnosed with CANDLE, Nakajo-Nishimura Syndrome (NNS), SAVI, AGS, or an equivalent syndrome, the need for previous biologic therapy is not required.
* Require treatment with oral corticosteroids (≥0.15 milligrams per kilogram per day [mg/kg/d] of prednisone or its equivalent) for control of systemic signs and symptoms of their chronic inflammatory disease for at least 2 weeks prior to study entry, or in the opinion of the investigator, have failed an adequate course of steroids. Treatment with or failure of treatment with steroids is not required for participants with AGS or a confirmed genetic diagnosis of CANDLE or SAVI.
* Have had previous documented elevations in acute-phase reactants (for example, high sensitivity C-reactive protein) considered to be the result of the inflammatory disease (participants with CANDLE or CANDLE-related conditions only).
* Have the ability to provide informed consent or have legal representative who is willing and able to provide written informed consent, provided that assent is obtained from participants at an age-appropriate level.

Exclusion Criteria:

* Have received an immunosuppressive biologic agent/monoclonal antibody within 4 half-lives prior to entry, for example, anakinra (4 half-lives=18 hours); etanercept (4 half-lives=18 days); infliximab; adalimumab (4 half-lives=36 days); use of intravenous immune globulin (IVIg) is permitted.
* Are pregnant or nursing at the time of entry.
* Are females of childbearing potential (women >12 or who have had at least 1 menstrual period regardless of age) who are sexually active and who do not agree to use 2 forms of highly effective methods of birth control or remain abstinent during the study and for at least 28 days following the last dose of investigational product.
* Are sexually active males who do not agree to use 2 forms of highly effective birth control with female partners of childbearing potential or remain abstinent during the study and for at least 28 days following the last dose of investigational product.
* Have had symptomatic herpes zoster infection within 12 weeks prior to entry or during the screening period.
* Have a history of disseminated/complicated herpes zoster (for example, multidermatomal involvement, ophthalmic zoster, central nervous system [CNS] involvement, postherpetic neuralgia).
* Have evidence of active infection, at the time of entry or during the screening period, that in the opinion of the investigator, would pose an unacceptable risk for participating in the study.
* Have a history of active hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV).
* Have documented high titer autoantibodies suggestive clinically of autoimmune diseases other than severe JDM.
* Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study.
* Have had a serious systemic or local infection (including an infectious mononucleosis-like illness or herpes zoster) within 12 weeks prior to entry or during the screening period.
* Have been exposed to a live vaccine within 12 weeks prior to entry or are expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study.

Note: Investigators should review the vaccination status of the participants and follow the local guidelines for vaccination with nonlive vaccines intended to prevent infectious disease prior to entering participants into the study.

* Have had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
* Have a serious and/or unstable illness that, in the opinion of the investigator, poses an unacceptable risk for the participant's participation in the study.
* Have an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine of <40 milliliters/minute/1.73 per square meter.
* Have or have had a history of lymphoproliferative disease; or signs or symptoms suggestive of possible lymphoproliferative disease, or active primary or recurrent malignant disease; or been in remission from clinically significant malignancy for <5 years.

Note: Participants with resolved cervical dysplasia, or no more than 3 successfully treated basal-cell carcinoma of the skin, may participate in this study.

* Have a history of chronic alcohol abuse or intravenous (IV) drug abuse within the 2 years prior to entry.
* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.
* Are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an investigational product or non-approved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Translational Autoinflammatory Disease (TADS), Bethesda, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Adang LA, Gavazzi F, D'Aiello R, Isaacs D, Bronner N, Arici ZS, Flores Z, Jan A, Scher C, Sherbini O, Behrens EM, Goldbach-Mansky R, Olson TS, Lambert MP, Sullivan KE, Teachey DT, Witmer C, Vanderver A, Shults J. Hematologic abnormalities in Aicardi Goutieres Syndrome. Mol Genet Metab. 2022 Aug;136(4):324-329. doi: 10.1016/j.ymgme.2022.06.003. Epub 2022 Jun 16. PMID 35786528
- [Derived] Kim H, Dill S, O'Brien M, Vian L, Li X, Manukyan M, Jain M, Adeojo LW, George J, Perez M, Grom AA, Sutter M, Feldman BM, Yao L, Millwood M, Brundidge A, Pichard DC, Cowen EW, Shi Y, Lu S, Tsai WL, Gadina M, Rider LG, Colbert RA. Janus kinase (JAK) inhibition with baricitinib in refractory juvenile dermatomyositis. Ann Rheum Dis. 2021 Mar;80(3):406-408. doi: 10.1136/annrheumdis-2020-218690. Epub 2020 Aug 25. No abstract available. PMID 32843325
- [Derived] Sanchez GAM, Reinhardt A, Ramsey S, Wittkowski H, Hashkes PJ, Berkun Y, Schalm S, Murias S, Dare JA, Brown D, Stone DL, Gao L, Klausmeier T, Foell D, de Jesus AA, Chapelle DC, Kim H, Dill S, Colbert RA, Failla L, Kost B, O'Brien M, Reynolds JC, Folio LR, Calvo KR, Paul SM, Weir N, Brofferio A, Soldatos A, Biancotto A, Cowen EW, Digiovanna JJ, Gadina M, Lipton AJ, Hadigan C, Holland SM, Fontana J, Alawad AS, Brown RJ, Rother KI, Heller T, Brooks KM, Kumar P, Brooks SR, Waldman M, Singh HK, Nickeleit V, Silk M, Prakash A, Janes JM, Ozen S, Wakim PG, Brogan PA, Macias WL, Goldbach-Mansky R. JAK1/2 inhibition with baricitinib in the treatment of autoinflammatory interferonopathies. J Clin Invest. 2018 Jul 2;128(7):3041-3052. doi: 10.1172/JCI98814. Epub 2018 Jun 11. PMID 29649002
- [Derived] Kim H, Brooks KM, Tang CC, Wakim P, Blake M, Brooks SR, Montealegre Sanchez GA, de Jesus AA, Huang Y, Tsai WL, Gadina M, Prakash A, Janes JM, Zhang X, Macias WL, Kumar P, Goldbach-Mansky R. Pharmacokinetics, Pharmacodynamics, and Proposed Dosing of the Oral JAK1 and JAK2 Inhibitor Baricitinib in Pediatric and Young Adult CANDLE and SAVI Patients. Clin Pharmacol Ther. 2018 Aug;104(2):364-373. doi: 10.1002/cpt.936. Epub 2017 Dec 8. PMID 29134648